CLINICAL TRIAL: NCT01205386
Title: Crosser Enters The Right Arterial Lumen
Acronym: CENTRAL
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: CR1055-01
Record Dates: First submitted 2010-04-26; First posted 2010-09-20 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Total Occlusion of Artery of the Extremities
Keywords: CTO; peripheral artery occlusive disease; PAOD; SFA; superficial femoral artery
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CROSSER
  Interventions: Device: 1. CROSSER System

INTERVENTIONS:
Device: 1. CROSSER System — The Crosser system will be used to recanalize the chronic total occlusion in the SFA (superficial femoral artery). The IVUS (Intravascular Ultrasound Imaging) System will be used in the treated occlusion after the Crosser to generate real-time images of the artery.
  Other Names: Crosser catheter; IVUS catheter

SUMMARY:
The purpose of this study is to determine if the CROSSER CTO Recanalization System can facilitate the successful crossing of Chronic Total Occlusions in the Central lumen of the Superficial Femoral Artery (SFA). A Chronic Total Occlusion (CTO) is defined as 100% narrowing of the artery, with no angiographically detectable antegrade blood flow, and the assessment that the lesion has been in existence for a minimum of 30 days. This study will enroll up to 100 patients at up to 8 clinical sites. The CROSSER CTO Recanalization System was cleared for commercialization by the US Food & Drug Administration. This study also involves an imaging device called the IVUS (Intravascular Ultrasound Imaging) catheter. This device has been cleared for commercialization by the US Food and Drug Administration and will be studied for its cleared intended use. The IVUS catheter is used to generate real-time images of the artery, which will allow for evaluation of the artery after the occlusion is crossed. This is a post-market registry.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have objective evidence of lower extremity ischemia and scheduled to undergo an endovascular recanalization.
* Occluded artery must be the native superficial femoral artery.
* Patient must have a totally occlusive lesion classified angiographically as absolute (100% occlusion with no flow).
* Patient's target vessel occlusion length is ≤ 30 cm.
* Patient's reference vessel diameter is greater than or equal to 3.0mm.
* Patient must be an acceptable candidate for PTA, peripheral artery bypass surgery or peripheral artery stent implantation.
* Female patients of child bearing potential must have a negative pregnancy test within 72 hours prior to the study procedure.
* Patient or guardian must have been informed of the nature of the study, agree to its provisions, and provide written informed consent.
* Patient is ≥ 18 years of age.

Exclusion Criteria:

* Patient has hypersensitivity or contraindication to aspirin, heparin or radiographic contrast agents which cannot be adequately pre-medicated.
* The patient requires immediate treatment in more than one occluded vessel, in any combination of grafts or native vessels.
* Patient's occlusion is a flush occlusion initiating less than 2cm from the ostium.
* Patient has planned infrainguinal intervention scheduled within 30 days after index procedure.
* The patient is currently participating in another investigational drug or device trial that may conflict with study data collection and has not completed the entire follow-up period.
* Patient has no collateral flow distal to the occlusion.
* Patient's target occlusion has a dissection that occurred within the past 60 days caused by a guidewire attempt.
* Patient has a history of bleeding diatheses, coagulopathy or will refuse blood transfusion in cases of emergency.
* Patient suffered recent (within the past 6 months) stroke or transient ischemic neurological attack (TIA).
* Patient suffered recent (within the past 6 months) significant gastrointestinal (GI) bleeding.
* Patient has other medical illnesses (i.e., cancer or congestive heart failure) that may cause the patient to be non-compliant with the protocol, confound the data interpretation or is associated with life-expectancy less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CTO who are indicated for recanalization.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Crosser navigates through the central lumen of the artery | At time of procedure (day 0)
  Successful navigation of the CROSSER CTO Recanalization Catheter in the central lumen of the artery as confirmed by Intravascular Ultrasound (IVUS) following recanalization

SECONDARY OUTCOMES:
Technical Success - crossing the CTO into the true distal lumen | At time of procedure (Day 0)
  The ability to facilitate crossing the CTO into the true distal lumen with the CROSSER Catheter and/or any conventional guidewire after use of the CROSSER.
Procedural Success - Technical success plus residual stenosis < 50% and improved flow | Time of Procedure (Day 0)
  Achievement of Technical Success plus a residual stenosis <50%, and improved flow verified angiographically, at the conclusion of the procedure.
Clinical Success - freedom from limb loss and repeat revascularization | 6 month follow-up
  Clinical Success - freedom from limb loss, and repeat revascularization (bypass surgery, or PTA) from index hospitalization through 6 moth follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P. Davis, MD, Principal Investigator — St. John Hospital & Medical Center
Locations (8):
- United States (8):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Mercy Heart and Vascular Center, Coon Rapids, Minnesota
  - Columbia University Medical Center, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Memphis Heart Clinic, Memphis, Tennessee